CLINICAL TRIAL: NCT02705651
Title: Non-functioning Pancreatic Neuroendocrine Tumors (NF-pNETs) in Multiple Endocrine Neoplasia Type 1 (MEN1) Treated With Somatostatin Analogs (SA) Versus NO Treatment - a Prospective, Randomized, Controlled Multicenter Study
Brief Title: Non-functioning Pancreatic Neuroendocrine Tumors in MEN1: Somatostatin Analogs Versus NO Treatment
Acronym: SANO
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Dr. Andreas Selberherr, M.D., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAN_001/16
Record Dates: First submitted 2016-03-02; First posted 2016-03-10 (Estimated); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Pancreatic Neuroendocrine Tumors in MEN1
MeSH Terms: interventions — CTAP octapeptide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Somatostatin-Analog (Experimental): A long acting somatostatin analog will be applied.
  Interventions: Drug: Somatostatin-Analog
- No treatment (No Intervention): This arm will be be the observational control according to the endpoints of the study. No intervention will be made.

INTERVENTIONS:
Drug: Somatostatin-Analog — A long-acting somatostatin-analog will be applied.
  Arms: Somatostatin-Analog

SUMMARY:
A.Background

More than 90% of patients with multiple endocrine neoplasia type 1 (MEN1) develop multiple pancreatic neuroendocrine tumors (pNETs). These tumors are the most common cause for premature death in MEN1.

While functioning pNETs must be treated to reduce or cure hormonal excess, the procedures for non-functioning pNETs are yet under discussion. Treatment ranges from watchful waiting to subtotal and total pancreatectomy. The latter may represent an "overtreatment", resulting in general complications and diabetic metabolic status.

The effect of somatostatin analogues (SAs) has shown promising results with regard to progression of non-functioning duodeno-pancreatic NETs. Treatment with SAs is highly safe and effective, resulting in long-time suppression of tumor growth.

B. Aim

In this study of MEN1 patients with non-functioning pNETs, the benefits of somatostatin analogs" (SAs; group 1) compared to "no treatment" (group 2) will be analyzed with regard to progression (tumor growth; development of new [functioning and non-functioning] neuroendocrine tumors and regional/distant metastasis).

C. Implementation

Patients will either receive Somatostatin Analogs (SAs) or no treatment. The observation period will be 60 months. The increase of tumor size and development of new tumors or metastasis will be monitored.

DETAILED DESCRIPTION:
1. Introduction

   1.1 Background

   Due to the genetic background of the disease, every single neuroendocrine cell of the pancreas is a potential progenitor of neuroendocrine tumors (NETs). More than 90% of patients with multiple endocrine neoplasia type 1 (MEN1) develop multiple pancreatic neuroendocrine tumors (pNETs) "viewable" by transgastric endosonography and/or cross sectional and/or functional imaging. These tumors are the most common cause for premature death in MEN1 (1, 2).

   While functioning pNETs are to be treated to reduce or cure hormonal excess, the strategies of addressing non-functioning (NF) pNETs are under discussion. Treatment ranges from "watchful waiting" to subtotal or total pancreatectomy (3-6). The latter may prove to be an "overtreatment" resulting in diabetic metabolic status and subsequently in general long-term complications.

   Somatostatin analogs (SAs) have shown promising results with regard to progression-free survival in patients with metastatic NETs of the midgut (9-11).

   As shown recently in a retrospective study of 40 patients with early-stage MEN1 duodeno-pancreatic NETs, treatment with SAs was safe and effective, resulting in long-time suppression of tumor and hormonal activity and 10% objective response. The authors suggest to start therapy with SAs early on in patients with MEN1-related NETs (12). Apart from this clinical study, there is one case report on SAs for MEN-1-related insulinoma (13).

   MEN1 is an orphan disease (ORPHA652).
2. Rationale and objectives

   In this prospective, randomized observation study, the benefits of subcutaneous application of somatostatin analogs (SAs) every 28 days (group 1) will be compared to no treatment (group 2). It has not been proven if the beneficial effects of SAs shown in advanced disease are also applicable to patients with early stage (≤20mm) pancreatic neuroendocrine tumors in MEN1. "Watch and wait" without medical treatment is the standard approach for MEN1 patients in this early stage of pancreatic disease. We hypothesize that SAs can decelerate tumor progression (according to our outcome parameters).
3. Study design

3.1 Design

Prospective, randomized, controlled, observation trial

3.2 Study population

Patients with proven MEN 1 (see eligibility criteria) will be recruited after discussing her/his individual clinical situation in the interdisciplinary tumor board.

The listed examinations and tests will be carried out in each patient before the first day of study participation:

* Medical history and physical examination
* Height and weight
* Biochemical parameters (chromogranin A [CgA] level)

3.3 Description of study days

The patients will be evaluated in six-monthly intervals biochemically and radiologically (according to the protocol below).

3.4 Withdrawal and replacement of subjects

Patients will be withdrawn under the following circumstances:

* At their own request
* If the investigators feel it would not be in the best interests of the patient to continue.

In all cases, the reasons why study subjects were withdrawn will be recorded in detail in the case report forms (CRFs) and in the subjects' medical records. Should the study be discontinued prematurely, all study materials (completed, partially completed and empty CRFs) will be retained.

4 Methods of evaluation

Functional imaging (DOTA-conjugated peptide PET-CT or MRI) will be performed and venous blood samples will be drawn as baseline evaluation for general laboratory tests and Chromogranin A (CgA).

4.1 Imaging modalities

DOTA-conjugated peptide PET-CT or MRI will be acquired on baseline and after 12, 24, 36, 48 and 60 months

Radiological interim assessments will be performed by MRI at 6, 18, 30, 42 and 54 months.

4.2 Laboratory parameters

A venous blood sample will be drawn at each assessment (baseline, 6, 12, 18, 24, 30, 36, 42, 48, 54, 60 months). CgA will be determined in each sample, general laboratory tests will be made yearly (starting from baseline).

4.3 Adverse events (AE)

An AE is any event during a clinical study, including intercurrent illness or accident, which impairs the well-being of the patient; it may also take the form of an abnormal laboratory value. The term AE does not imply a causal relationship with the study therapy.

All subjects experiencing AEs - whether considered associated with the study therapy or not - will be monitored until symptoms subside and any abnormal laboratory values have returned to baseline, or until there is a satisfactory explanation for the changes observed, or until death, in which case a full pathologist's report will be supplied, if possible. All findings must be reported on an "AE" page in the "case report form (CRF)".

All AEs are divided into the categories "serious" and "non-serious". This determines the procedure that must be used to report/document the AE (see below).

4.3.1 Definition of serious and non-serious adverse events

A serious AE is:

* Any event that is fatal or life-threatening
* Any event that is permanently disabling
* Any event that requires hospitalization AEs that do not fall into these categories are defined as non-serious.

4.3.2 Reporting /documentation of adverse events AEs will be collected by spontaneous reporting.

4.3.3 Assessment of severity

Regardless of the classification of an AE as serious or non-serious (see above), its severity must be assessed as mild, moderate or severe, according to medical criteria alone:

Mild = does not interfere with routine activities, considered as acceptable

Moderate = interferes with routine activities

Severe = impossible to perform routine activities, considered as unacceptable

Further categories: Requires treatment, requires discontinuation of study, or has residual effect.

It should be noted that a severe AE need not be serious in nature and that a serious AE need not, by definition, be severe.

Regardless of severity, all serious AEs must be reported as above.

4.4 Data handling procedures A CRF will be completed for each patient. Trained personnel will check the entries and any errors or inconsistencies will be clarified immediately. The results of the pre-study screening examination will be documented in the study master file.

4.5 Biometric methods

4.5.1 Biometric methods

1. Descriptive analysis
2. After analysis for data distribution, parametric or non-parametric statistical tests will be applied

4.5.2 Biometric methods - adverse events/safety investigations

All AEs will be properly listed and an appropriate method will be used to summarize the data.

5 Ethical and legal aspects The study will be performed in accordance with the guidelines of the Declaration of Helsinki (1964), including current revisions.

5.1 Informed consent of the patient Before being admitted to the clinical investigation, patients must have consented to participate after the nature, scope and possible consequences of the clinical study have been made understandable to them in writing.

Patients must give a written consent. Their consent will be confirmed by the signature of one investigator.

5.2 Acknowledgment/approval of the study Before the start of the study, the study protocol will be submitted to the Ethics Committee of the Medical University of Vienna and, if necessary, to the responsible Ethics Committees of the participating centers.

5.3 Confidentiality

All subjects' names will be kept secret in the investigators' files. Subjects will be identified throughout documentation and evaluation by the number allotted to them at the beginning of the study. The subjects will be informed that all study findings will be stored and handled in strictest confidence.

6 Documentation and use of study findings

6.1 Documentation of study findings All findings collected during the study will be entered on the CRFs. CRFs will be completed immediately after the final examination.

6.2 Use of study findings The findings of this study will be published by the investigators in a scientific journal and presented at scientific meetings. The manuscript will be circulated to all co-investigators before submission.

7 Protocol amendments If any modifications become necessary or desirable, these will be documented in writing; major changes will require the approval of all investigators and the Ethics Committee.

ELIGIBILITY:
Inclusion Criteria:

* Verified MEN1 syndrome by molecular genetics (known mutation)
* Non-functioning pNET
* Largest ("leading") pancreatic tumor with ≤20 mm in diameter and (if present) one small tumor <15 mm in diameter as reference lesion
* G1 or G2 (Ki-67 ≤ 10%) according to endoscopic ultrasound/fine-needle aspiration (EUS/FNA) acquired by 19-gauge needle
* Functional imaging: Ga68-DOTA-conjugated peptide positron emission tomography (PET) computed tomography (CT) or preferably Ga68-DOTA-conjugated peptide magnetic resonance imaging (MRI)
* Tumor(s) limited to the pancreas (N0, M0)

Exclusion Criteria:

* Functioning tumor - hormone excess
* Neuroendocrine carcinoma (G3)
* Metastatic disease (N1, M1)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2019-12 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Growth rate of the tumor in mm | 5 years
  The growth rate of the leading lesion (≥20mm in diameter) will be radiologically controlled in six-monthly intervals. Growth rate will be compared between the groups.

SECONDARY OUTCOMES:
Documentation of new tumors | 5 years
  In intervals of 6 months radiologic examinations of the pancreas will be made, thereby newly developed tumors can be documented and will be compared between the groups.
Documentation of lymph node and/or distant metastases | 5 years
  Functional imaging will be made in intervals of 12 months. With this modality newly arisen metastatic lesions can be documented. The development of those lesions will be compared between the groups.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Selberherr, M.D., Principal Investigator — Medical University of Vienna

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dean PG, van Heerden JA, Farley DR, Thompson GB, Grant CS, Harmsen WS, Ilstrup DM. Are patients with multiple endocrine neoplasia type I prone to premature death? World J Surg. 2000 Nov;24(11):1437-41. doi: 10.1007/s002680010237. PMID 11038219
- [Background] Ito T, Igarashi H, Uehara H, Berna MJ, Jensen RT. Causes of death and prognostic factors in multiple endocrine neoplasia type 1: a prospective study: comparison of 106 MEN1/Zollinger-Ellison syndrome patients with 1613 literature MEN1 patients with or without pancreatic endocrine tumors. Medicine (Baltimore). 2013 May;92(3):135-181. doi: 10.1097/MD.0b013e3182954af1. PMID 23645327
- [Background] Doherty GM, Thompson NW. Multiple endocrine neoplasia type 1: duodenopancreatic tumours. J Intern Med. 2003 Jun;253(6):590-8. doi: 10.1046/j.1365-2796.2003.01163.x. PMID 12755954
- [Background] Gauger PG, Thompson NW. Early surgical intervention and strategy in patients with multiple endocrine neoplasia type 1. Best Pract Res Clin Endocrinol Metab. 2001 Jun;15(2):213-23. doi: 10.1053/beem.2001.0136. PMID 11472035
- [Background] Kouvaraki MA, Shapiro SE, Cote GJ, Lee JE, Yao JC, Waguespack SG, Gagel RF, Evans DB, Perrier ND. Management of pancreatic endocrine tumors in multiple endocrine neoplasia type 1. World J Surg. 2006 May;30(5):643-53. doi: 10.1007/s00268-006-0360-y. PMID 16680581
- [Background] Akerstrom G, Hessman O, Skogseid B. Timing and extent of surgery in symptomatic and asymptomatic neuroendocrine tumors of the pancreas in MEN 1. Langenbecks Arch Surg. 2002 Mar;386(8):558-69. doi: 10.1007/s00423-001-0274-6. Epub 2002 Jan 24. PMID 11914931
- [Background] Gauger PG, Doherty GM, Broome JT, Miller BS, Thompson NW. Completion pancreatectomy and duodenectomy for recurrent MEN-1 pancreaticoduodenal endocrine neoplasms. Surgery. 2009 Oct;146(4):801-6; discussion 807-8. doi: 10.1016/j.surg.2009.06.038. PMID 19789041
- [Background] Adkisson CD, Stauffer JA, Bowers SP, Raimondo M, Wallace MB, Riegert-Johnson DL, Asbun HJ. What extent of pancreatic resection do patients with MEN-1 require? JOP. 2012 Jul 10;13(4):402-8. doi: 10.6092/1590-8577/657. PMID 22797396
- [Background] Rinke A, Muller HH, Schade-Brittinger C, Klose KJ, Barth P, Wied M, Mayer C, Aminossadati B, Pape UF, Blaker M, Harder J, Arnold C, Gress T, Arnold R; PROMID Study Group. Placebo-controlled, double-blind, prospective, randomized study on the effect of octreotide LAR in the control of tumor growth in patients with metastatic neuroendocrine midgut tumors: a report from the PROMID Study Group. J Clin Oncol. 2009 Oct 1;27(28):4656-63. doi: 10.1200/JCO.2009.22.8510. Epub 2009 Aug 24. PMID 19704057
- [Background] Caplin ME, Pavel M, Cwikla JB, Phan AT, Raderer M, Sedlackova E, Cadiot G, Wolin EM, Capdevila J, Wall L, Rindi G, Langley A, Martinez S, Blumberg J, Ruszniewski P; CLARINET Investigators. Lanreotide in metastatic enteropancreatic neuroendocrine tumors. N Engl J Med. 2014 Jul 17;371(3):224-33. doi: 10.1056/NEJMoa1316158. PMID 25014687
- [Background] Faiss S, Pape UF, Bohmig M, Dorffel Y, Mansmann U, Golder W, Riecken EO, Wiedenmann B; International Lanreotide and Interferon Alfa Study Group. Prospective, randomized, multicenter trial on the antiproliferative effect of lanreotide, interferon alfa, and their combination for therapy of metastatic neuroendocrine gastroenteropancreatic tumors--the International Lanreotide and Interferon Alfa Study Group. J Clin Oncol. 2003 Jul 15;21(14):2689-96. doi: 10.1200/JCO.2003.12.142. PMID 12860945
- [Background] Ramundo V, Del Prete M, Marotta V, Marciello F, Camera L, Napolitano V, De Luca L, Circelli L, Colantuoni V, Di Sarno A, Carratu AC, de Luca di Roseto C, Colao A, Faggiano A; Multidisciplinary Group for Neuroendocrine Tumors of Naples. Impact of long-acting octreotide in patients with early-stage MEN1-related duodeno-pancreatic neuroendocrine tumours. Clin Endocrinol (Oxf). 2014 Jun;80(6):850-5. doi: 10.1111/cen.12411. Epub 2014 Feb 19. PMID 24443791
- [Background] Marciello F, Di Somma C, Del Prete M, Marotta V, Ramundo V, Carratu A, de Luca di Roseto C, Camera L, Colao A, Faggiano A. Combined biological therapy with lanreotide autogel and cabergoline in the treatment of MEN-1-related insulinomas. Endocrine. 2014 Aug;46(3):678-81. doi: 10.1007/s12020-013-0145-2. Epub 2014 Jan 3. PMID 24385268